CLINICAL TRIAL: NCT05625789
Title: How to Get Started: Identifying the Critical Ingredients to Improve Gait Initiation in Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: LSVT Global (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 22-2628
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease
Keywords: Freezing of Gait; Gait Initiation
MeSH Terms: conditions — Parkinson Disease | interventions — Postural Balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postural control (weight shifting) training followed by steady state gait training. (Experimental): For postural control training, participants will be provided visual biofeedback to increase weight shift prior to the first step. The feedback program cues participants to reach a target amount of weight shift. Once the target is reached, participants are cued to initiate walking. Participants will complete a total of 30 minutes of training, ensuring at least 45 repetitions.
  To create larger amplitude movements during steady state gait, participants will walk on a treadmill set to their comfortable gait speed while attempting to match their steps to a metronome beeping at 85% of their comfortable cadence. Participants will complete a total of 10 minutes of treadmill walking with rest breaks as needed. Next, participants will walk overground to a metronome beeping at 115% of their comfortable cadence with a goal of 10 total minutes of training.
  Each training will be three times per week for two weeks. There is a one week break between the two trainings.
  Interventions: Behavioral: Postural control (weight shift) training; Behavioral: Steady state gait training
- Steady state gait training followed by postural control (weight shifting) training. (Experimental): To create larger amplitude movements during steady state gait, participants will walk on a treadmill set to their comfortable gait speed while attempting to match their steps to a metronome beeping at 85% of their comfortable cadence. Participants will complete a total of 10 minutes of treadmill walking with rest breaks as needed. Next, participants will walk overground to a metronome beeping at 115% of their comfortable cadence with a goal of 10 total minutes of training.
  For postural control training, participants will be provided visual biofeedback to increase weight shift prior to the first step. The feedback program cues participants to reach a target amount of weight shift. Once the target is reached, participants are cued to initiate walking. Participants will complete a total of 30 minutes of training, ensuring at least 45 repetitions.
  Each training will be three times per week for two weeks. There is a one week break between the two trainings.
  Interventions: Behavioral: Postural control (weight shift) training; Behavioral: Steady state gait training

INTERVENTIONS:
Behavioral: Postural control (weight shift) training — Visual cues to improve amplitude of weight shift prior to initiating gait.
Behavioral: Steady state gait training — Auditory cues are provided to increase amplitude of movement (e.g., step length) during continuous walking, to determine its effects on gait initiation amplitude of movement.

SUMMARY:
The purpose of this study is to understand the treatment approach (i.e., targeting gait or targeting the postural adjustment prior to gait) that is most effective at improving gait initiation dynamics in people with Parkinson disease. Ten adults with idiopathic Parkinson disease who self-report difficulty initiating gait will complete the study. The investigators will be using a randomized crossover design, where the participants will participate in two series of training (i.e., postural training and steady-state gait training) with a one-week washout between trainings. Investigators will evaluate the changes induced in gait initiation postural adjustment size, first step length, and first step speed from each intervention. Due to the anticipated limitation of steady-state walking to directly address postural adjustment amplitude, it is hypothesized that training for larger amplitude weight shift during gait initiation will yield improved gait initiation dynamics compared to training with large amplitude movements during steady-state walking.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson disease characterized by asymmetrical onset of at least 2 of 3 cardinal signs (resting tremor, bradykinesia, or rigidity) with no atypical signs or exposure to dopamine-blocking drugs
* The presence of mild to moderate gait or balance impairment (a rating of 1-2 on MDS Unified Parkinson Disease Rating Scale (MDS-UPDRS) item 10 [gait] or rating 1-3 on item 12 [postural stability]
* Hoehn & Yahr stages 1-3 ("on" for those who fluctuate)
* Self-report of difficulty with freezing of gait (i.e., a rating of 1-4 on question 3 of the Freezing of Gait Questionnaire)
* All participants must be able to walk > 5 minutes at greater than or equal to 80% of comfortable gait speed (CGS) on the treadmill and > 5 minutes over ground without assistance or an assistive device.

Exclusion Criteria:

* Uncontrolled cardiorespiratory/metabolic disease, vestibular dysfunction that may affect gait or balance
* Parkinson's related or unrelated dementia (i.e. Montreal Cognitive Assessment score <21)
* Comfortable over ground walking speed of less than 0.5m/s
* History of traumatic brain injury
* self-reported deafness or blindness as this would impair the patient's ability to hear cues or ambulate safely within the lab environment
* other neurological disorders or orthopedic injury that may affect gait
* recent orthopedic surgery (in the last 6 months)
* Participants will also be excluded if they have severe communication impairments, which could impede understanding of the purpose or procedures of the study or an inability to comply with experimental procedures
* Participants who are currently receiving supervised physical therapy services

Ages: 35 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
Change in First Step Length from Baseline to Conclusion of the first block of training | Baseline, at the conclusion of the first block of training (approximately 2 weeks)
  Length of the first step during gait initiation (i.e., distance from stepping limb heel marker at quiet stance to heel marker of stepping limb at heel strike of the first step forward).
Change in First Step Length from end of first block of training to training 2 pre-test | Conclusion of first training block, just prior to beginning the second training series (1 week)
  Length of the first step during gait initiation (i.e., distance from stepping limb heel marker at quiet stance to heel marker of stepping limb at heel strike of the first step forward).
Change in First Step Length from training block 2 pre-test to conclusion of second block of training | Prior to beginning second block of training, at the conclusion of second block of training (2 weeks)
  Length of the first step during gait initiation (i.e., distance from stepping limb heel marker at quiet stance to heel marker of stepping limb at heel strike of the first step forward).
Change in First Step Length from conclusion of second training block to 1 week follow up from second training block | Conclusion of second training block, 1 week follow up from conclusion of second training block (1 week)
  Length of the first step during gait initiation (i.e., distance from stepping limb heel marker at quiet stance to heel marker of stepping limb at heel strike of the first step forward).

SECONDARY OUTCOMES:
Change in Mediolateral Anticipatory Postural Adjustment (APA) Size from Baseline to Conclusion of the first block of training | Baseline, at the conclusion of the first block of training (approximately 2 weeks)
  Center of pressure displacement towards the stepping limb from quiet stance until toe off of the stepping limp (i.e., the initiation of gait).
Change in Mediolateral Anticipatory Postural Adjustment (APA) Size from end of first block of training to training 2 pre-test | Conclusion of first training block, just prior to beginning the second training series (1 week)
  Center of pressure displacement towards the stepping limb from quiet stance until toe off of the stepping limp (i.e., the initiation of gait).
Change in Mediolateral Anticipatory Postural Adjustment (APA) Size from training block 2 pre-test to conclusion of second block of training | Prior to beginning second block of training, at the conclusion of second block of training (2 weeks)
  Center of pressure displacement towards the stepping limb from quiet stance until toe off of the stepping limp (i.e., the initiation of gait).
Change in Mediolateral Anticipatory Postural Adjustment (APA) Size from conclusion of second training block to 1 week follow up from second training block | Conclusion of second training block, 1 week follow up from conclusion of second training block (1 week)
  Center of pressure displacement towards the stepping limb from quiet stance until toe off of the stepping limp (i.e., the initiation of gait).
Change in First Step Speed from Baseline to Conclusion of the first block of training | Baseline, at the conclusion of the first block of training (approximately 2 weeks)
  First step speed is measured by dividing the first step length by the time it takes to take the first step - which is calculated as the time from toe off of the stepping limb to heel strike of the stepping limb.
Change in First Step Speed from end of first block of training to training 2 pre-test | Conclusion of first training block, just prior to beginning the second training series (1 week)
  First step speed is measured by dividing the first step length by the time it takes to take the first step - which is calculated as the time from toe off of the stepping limb to heel strike of the stepping limb.
Change in First Step Speed from training block 2 pre-test to conclusion of second block of training | Prior to beginning second block of training, at the conclusion of second block of training (2 weeks)
  First step speed is measured by dividing the first step length by the time it takes to take the first step - which is calculated as the time from toe off of the stepping limb to heel strike of the stepping limb.
Change in First Step Speed from from conclusion of second training block to 1 week follow up from second training block | Conclusion of second training block, 1 week follow up from conclusion of second training block (1 week)
  First step speed is measured by dividing the first step length by the time it takes to take the first step - which is calculated as the time from toe off of the stepping limb to heel strike of the stepping limb.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lewek, PhD, Study Director — UNC Chapel Hill; Chelsea P Duppen, DPT, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning after publication to five years following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill.
Time Frame: Results will be shared following publication and up to five years following publication.
Access Criteria: The investigator who proposes to use the data must have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and must execute a data use/sharing agreement with the University of North Carolina at Chapel Hill.